Title: Effect of Different Plane Blocks on Quality of Recovery and Postoperative Pain After

Laparoscopic Hysterectomy

**Protocol ID: 2022/12** 

ClinicalTrials.gov ID: NCT05780333

Document Date: 21.01.2023 / Version 1

**Informed Consent Form (ICF)** 

**Active Arm (ESP Block)** 

This study is a research study.

Purpose of the Study: After each surgery, patients feel pain at different rates depending on

the type of surgery. This pain is tried to be minimized with painkillers given orally and

intravenously. In recent years, in order to protect against the side effects of these given

painkillers and to reduce pain more effectively, needle procedures are performed before

waking up from the surgery and the nerves that perceive the pain are anesthetized. In order to

minimize the pain felt after closed uterus removal operations, there are two different pain

relief needle procedures that can be applied in the usual situation. There is scientific data

showing that both processes are beneficial. Both methods have been used for a long time to

reduce pain. This study is a scientific research conducted for the purpose of comparing two

different pain relief procedures currently applied, in which no additional procedures were

performed.

Method of the Study: This study will be carried out at Mentese State Hospital. You will be

asked to fill out a questionnaire on your quality of life before and at the 24th hour after the

surgery, and to express the severity of your pain during the 24 hours you stay in the hospital.

Participation in the study is on a voluntary basis. It is planned to include volunteer patients

who had closed uterine removal surgery within a six (6) month period.

Both procedures are the method of administering drugs that numb the nerves between the

muscles (the pain-sensing nerves pass through this muscle group). The difference between

them is that one transaction is made from the profit, while the other is done from the back.

The procedure that will be applied to you is the type of operation applied from the back. The

procedures are applied with the help of a thin needle, which is applied just before waking up

when the surgery is over and lasts for 5-10 minutes. In the procedures, the right place will be determined by ultrasound and the nerve endings that detect the pain will be temporarily anesthetized. Even if you do not participate in the study, these procedures are performed by your anesthesiologist to manage post-operative pain. Which of the procedures to be performed is determined with the help of a computer program, and your comfort will increase after the operation, no matter which procedure is applied.

It is your responsibility to read, understand and fill out the questionnaires given to you regarding this research, and to give a number between 1 and 10 (1: I have no pain, 10: the most severe pain I have ever heard in my life) when asked about your pain status. All your medical and identity information will be kept confidential, even if the research is published, your identity information will not be given. You can access your own medical information whenever you want.

Participation in this research is entirely at your own discretion. You can refuse to participate in the research or leave the research at any stage; this will in no way damage the relationship of trust between you and your doctor and will not interrupt your follow-up process.

## Name / Surname / Telephone of the Person Who Can Be Reached 24 Hours During the Research:

Volunteers can contact MD. Pelin DILSIZ EKER at +905378401872 to obtain information about their rights.

## **Volunteer Statement:**

I have read and verbally listened to the above information that should be given to the volunteer before starting the research. Written and verbal explanation about the research whose subject and purpose is stated above was given to me by MD. Pelin DILSIZ EKER. I asked all the questions that came to my mind to the researcher, and I understood in detail all the written and verbal explanations made to me. I was given sufficient time to decide whether I wanted to participate in the study. I know that I have voluntarily participated in the research and that I can leave the research at any time with or without justification. I agree to participate in the research in question voluntarily without any pressure or coercion, I authorize the

research director to review my medical information, and I voluntarily accept the invitation to participate in the research in question without any coercion or pressure.

| Volunteer: |
|-----------------|
| Name – Surname: |
| Date: |
| Signature: |

## **Principal Investigator:**

MD. Pelin DILSIZ EKER

Mentese State Hospital, Department of Anesthesiology and Reanimation

Number: +905378401872